CLINICAL TRIAL: NCT04611620
Title: Biobehavioral Correlates of Cancer-related Cognitive Dysfunction and Its Co-occurring Symptoms
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Diane Von Ah, Associate Dean of Academic Operations, Indiana University
Other Study IDs: NURS-IIR-IUSCCC-0748
Record Dates: First submitted 2020-10-12; First posted 2020-11-02 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Survivorship; Cognitive Dysfunction; Pain; Depression; Anxiety; Fatigue; Sleep Disturbance
Keywords: Breast Cancer and Colorectal Cancer; Co-Occurring Symptoms
MeSH Terms: conditions — Cognitive Dysfunction; Pain; Depression; Anxiety Disorders; Fatigue; Parasomnias; Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The NIH NINR lab will run genome-wide sequencing per an approved and standardized protocol. In this study, we will focus on 3 genetic SNP variants of BDNF, APOE, and COMT (described previously). After final batch analyses, only outcome data with the unique identification numbers will be transferred via secure server to be linked back with the other survey and neuropsychological data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer and Colorectal Cancer Survivors: The purpose of this study is to explore the factors related with cognitive concerns and other symptoms in breast and colorectal cancer survivors.
  Interventions: Behavioral: Cognitive Dysfunction

INTERVENTIONS:
Behavioral: Cognitive Dysfunction — To fully characterize factors associated with cognitive dysfunction in BCS and CRC survivors that have cognitive concerns and (2) to fully characterize factors associated with psychoneurological symptom cluster in BCS and CRC survivors.

SUMMARY:
This descriptive, cross-sectional study will evaulate and fully characterize factors associated with cognitive dysfunction in Breast Cancer (BCS) and Colorectal Cancer (CRC) survivors that have cognitive concerns, and factors associated with psychoneurological symptom cluster in BCS and CRC survivors.

DETAILED DESCRIPTION:
Primary Aim: To identify demographic factors (age and education), medical and cancer treatment-related factors (comorbidities and treatment type), psychosocial factors (perceived stress, affect, optimism, coping, emotional support), cancer-related symptoms (pain, depression, anxiety, fatigue and sleep disturbance), and genetic factors (APOE, COMT, BDNF) associated with the level of subjective or the level of objective cognitive dysfunction in breast cancer and colorectal cancer survivors.

Secondary Aim: To identify demographic factors (age and education), medical and cancer treatment-related factors (comorbidities and treatment type), psychosocial factors (perceived stress, affect, optimism, coping, emotional support), and genetic factors (APOE, COMT, BDNF) associated with psychoneurological symptom cluster using either subjective or objective cognitive dysfunction in breast cancer and colorectal cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Breast cancer survivors:

1. Female BCS
2. ≥ 21 years of age and older
3. Ability to provide written consent and HIPAA authorization
4. ≥6 months post-adjuvant therapy and neo-adjuvant therapy for early stage (Stage I-IIIA) breast cancer.

   Current Aromatase Inhibitors or Tamoxifen treatment at time of enrollment is allowed.
5. Identify cognitive concerns (select yes)

Inclusion Criteria for Colorectal cancer survivors:

1. Male or female CRC survivors
2. Ability to provide written consent and HIPAA authorization
3. ≥ 21 years of age and older
4. ≥6 months post-adjuvant therapy and neo-adjuvant therapy for early stage (stage I-III) CRC
5. Identify cognitive concerns (select yes)

Exclusion Criteria:

1. Report metastatic breast or colorectal cancer (Stage IV) at time of consenting.
2. Unable to read and understand English to complete survey questionnaires.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 465 breast and colorectal cancer patients will be recruited for this study. Breast and colorectal cancer survivors.
  The eligibility checklist is a self-report questionnaire. Participants will be asked to self-identify that they are 21 years of age or older, had been diagnosed with breast or colorectal cancer excluding Stage IV (those without distant metastasis) and have completed treatment (adjuvant or neo-adjuvant) at least 6 months prior to completing the survey. In addition, as part of the eligibility checklist, participants will need to self-rate that they have cognitive concerns (select yes).
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Subjective Cognitive Dysfunction | greater than or equal to 6 months post cancer treatment
  PROMIS - Cognitive Abilities and Concerns

SECONDARY OUTCOMES:
Objective Cognitive Dysfunction | greater than or equal to 6 months post cancer treatment
  Visual Episodic Memory
Objective Cognitive Dysfunction | greater than or equal to 6 months post cancer treatment
  Working Memory
Objective Cognitive Dysfunction | greater than or equal to 6 months post cancer treatment
  Executive Functioning
Objective Cognitive Dysfunction | greater than or equal to 6 months post cancer treatment
  Sustained Attention
Objective Cognitive Dysfunction | greater than or equal to 6 months post cancer treatment
  Visuospatial Working Memory

CONTACTS AND LOCATIONS:
Overall Officials: Diane Von Ah, PhD, Principal Investigator — IU
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Goto T, Saligan LN, Li X, Xiang L, Kwiat C, Nguyen C, Crouch A, Von Ah D. Associations of brain-derived neurotrophic factor rs6265 polymorphism and cognitive function in breast cancer survivors from a cross-sectional study. Cancer Med. 2024 Jan;13(2):e6975. doi: 10.1002/cam4.6975. PMID 38379321
- [Derived] Storey S, Draucker C, Haunert L, Von Ah D. The Experience of Peripheral Neuropathy Symptoms in Breast Cancer Survivors With Diabetes. Cancer Nurs. 2024 Jul-Aug 01;47(4):E279-E286. doi: 10.1097/NCC.0000000000001253. Epub 2023 May 26. PMID 37232534